CLINICAL TRIAL: NCT04562987
Title: The Patterns of Activity and Cognition During Treatment (PACT) Study
Acronym: PACT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nebraska (Other)
Collaborators: National Institute of General Medical Sciences (NIGMS) (NIH); Wake Forest University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Supportive Care
Other Study IDs: 0736-19-FB; 1U54GM115458 (NIH)
Record Dates: First submitted 2020-09-09; First posted 2020-09-24 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Breast Neoplasms; Breast Cancer Female
Keywords: breast cancer; physical activity; cognition; chemotherapy
MeSH Terms: conditions — Breast Neoplasms; Motor Activity | interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Core Component (tele-coaching, emails, smartphone app & Fitbit) (Active Comparator): All participants will receive the Core component, which includes access to weekly tele-coaching, weekly emails from the interventionist, a smartphone app, and a Fitbit monitor. Tele-coaching will include discussion of general cancer-related and wellness topics, and the smartphone app will have basic activity monitoring features.
  Interventions: Behavioral: Attentional Control
- Move (tele-coaching calls, smartphone app & Move goals & badges) (Experimental): Tele-coaching calls for Move participants will be based in social cognitive theory to encourage behavior adoption and goal setting focused on reducing prolonged sitting. Smartphone app features include activity monitoring that visualizes progress toward Move-based goals and goal achievement badges specific to Move.
  Interventions: Behavioral: Physical Activity
- Exercise (tele-coaching calls & smartphone app) (Experimental): Tele-coaching calls for Exercise participants will be based in social cognitive theory to encourage behavior adoption and goal setting focused on engaging in 30 minutes of moderate-intensity physical activity per day (in 10+ minute bouts). Smartphone app features include activity monitoring that visualizes progress toward Exercise-based goals and goal achievement badges specific to Exercise.
  Interventions: Behavioral: Physical Activity
- Combo (Move+Exercise) (Experimental): Includes tele-coaching that encourages behavior adoption and goal setting focused on reducing prolonged sitting and engaging in 30+ minutes of physical activity per day. Participants are able to visualize progress toward Move and Exercise goals and are eligible to receive achievement badges for Move and Exercise.
  Interventions: Behavioral: Physical Activity

INTERVENTIONS:
Behavioral: Physical Activity — Mobile app intervention delivered during chemotherapy for breast cancer that combines goal setting, behavioral monitoring, and goal achievement badges with telecoaching to achieve physical activity prescriptions.
  Arms: Combo (Move+Exercise); Exercise (tele-coaching calls & smartphone app); Move (tele-coaching calls, smartphone app & Move goals & badges)
Behavioral: Attentional Control — Mobile app intervention delivered during chemotherapy for breast cancer that includes telecoaching on general and cancer-related health topics and basic physical activity monitoring.
  Arms: Core Component (tele-coaching, emails, smartphone app & Fitbit)

SUMMARY:
Aim 1: This pilot study tests the feasibility and acceptability of a mobile app-based behavioral intervention in 40 women receiving chemotherapy for breast cancer. Participants will be randomized to receive app components following a 2x2 factorial design. Feasibility will be assessed by participant recruitment yield, intervention adherence, contamination, and retention. Acceptability will be assessed by participant ratings and perceptions of intervention components as measured at post-intervention (1 month post-chemotherapy).

Aim 2: Examine preliminary efficacy of the intervention components (i.e., Move, Exercise, Core) delivered alone (i.e., main effects) and in combination (i.e., interaction effects; Move+Exercise) on executive function and working memory at post-intervention. These data will inform the sample size needed for a fully-powered randomized controlled trial. Aim 2 outcomes will be measured at pre-intervention (before the first or second chemotherapy cycle) and post-intervention, and include accelerometry and neurocognitive testing.

Exploratory Aim: Explore the effects of the intervention components on correlates of cancer-associated cognitive decline. Exploratory outcomes will be measured at pre- and post-intervention and include patient-reported outcomes, specifically cancer-related fatigue. Participants will also completed brief ecological momentary assessments (EMAs) their mobile phones across four 14-day measurement bursts at pre-intervention, mid-chemotherapy, and 1 month post-chemotherapy to further explore associations among behavioral patterns, cognition, and correlates.

DETAILED DESCRIPTION:
Cancer-related cognitive impairment (CRCI) is a research priority due to its rising prevalence and dramatic impacts on survivors' quality of life and health long-term. Strong evidence supports the efficacy of physical activity (PA) for improving cognitive function and key CRCI correlates. The aim of the proposed study is to pilot test an innovative, mHealth intervention designed to ameliorate CRCI in women receiving chemotherapy for breast cancer. This study will employ an efficient 2x2 factorial design to compare PA prescriptions targeting frequent PA of any intensity and reduced daily sitting (Move); aerobic exercise (consistent with PA guidelines for cancer survivors; Exercise); both (Move+Exercise); or none (Core). The main and interactive effects of these intervention components on CRCI and its underlying mechanisms will be tested across the breast cancer trajectory. Aim 1: This pilot study aims to test the feasibility and acceptability of the mHealth intervention in 40 women receiving chemotherapy for breast cancer. Feasibility will be assessed by participant recruitment yield, intervention adherence, contamination, and retention. Acceptability will be assessed by participant ratings and perceptions of intervention components as measured at a baseline orientation and at post-intervention (1 month post-chemotherapy). Aim 2: Examine preliminary efficacy of the intervention components (i.e., Move, Exercise, Core) delivered alone (i.e., main effects) and in combination (i.e., interaction effects) on executive function and working memory at post-intervention. These data will inform the sample size needed for a fully-powered randomized controlled trial. Aim 2 outcomes will be measured at pre-intervention (before the first or second chemotherapy cycle) and post-intervention, and include accelerometry and neurocognitive testing. Exploratory Aim: Explore the effects of the intervention components on CRCI correlates. Exploratory outcomes will be measured at pre- and post-intervention and include patient-reported outcomes (e.g., fatigue, depressive symptoms). Participants will also complete brief ecological momentary assessments (EMAs) on their mobile phones across four 14-day measurement bursts to further explore associations among behavioral patterns, cognition, and CRCI correlates. To test the specific aims, women diagnosed with breast cancer and scheduled to receive 3-6 months of chemotherapy (N=40) will be randomized to receive select mHealth intervention components, including Core (attentional control), Move, Exercise, or Move+Exercise (n=10 each condition). Data will be analyzed using descriptive statistics and axial coding (Aim 1); analysis of covariance and standard mean difference (Aim 2 and Exploratory); and hierarchical linear modeling (Exploratory). Findings will provide the necessary pilot data to support a grant application for a fully-powered trial.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Aged 21 years or older
* First, primary diagnosis of Stage I-III breast cancer
* Scheduled to receive chemotherapy for 3-6 months. While evidence suggests declines in cognition and brain health due to cancer may be evident both in women who receive and who do not receive chemotherapy, those receiving chemotherapy consistently experience the greatest changes.
* Has received no more than one cycle of chemotherapy
* Agree to be randomized to one of the intervention components
* Owns an Android or iPhone smartphone
* Fitbit specific criteria:

  * Compatible mobile device, laptop computer, or desktop computer
  * Willingness to continuously wear the Fitbit device during waking hours for the duration of the study period. Individuals not willing to wear the Fitbit during sleep will be eligible to participate.
  * Willingness and ability to charge the Fitbit device at home every 3-4 days and synchronize the Fitbit device multiple times daily.
* English reading and speaking
* Receive physician's clearance to participate in an exercise program
* Provide written informed consent to participate in the study
* No history or evidence of dementia (score >21 on the Modified Telephone Interview for Cognitive Status [TICS-M].73

Exclusion Criteria:

* Males. Breast cancer is often classified specifically as female breast cancer, as 99% of cases occur in women. Our small sample size does not statistically justify the inclusion of males in this study. As such, only female subjects will be included in this research
* Is scheduled to receive <3 months or >6 months of chemotherapy
* Has received 2+ cycles of chemotherapy at enrollment
* Stage 0 breast cancer diagnosis or metastatic disease
* Second cancer diagnosis (excluding non-invasive skin cancers; including breast cancer recurrence)
* Is not cleared to participate in exercise by a physician.
* Unwilling to complete baseline behavioral, neurocognitive, and patient-reported assessments (accelerometry, cognitive tasks, questionnaires)
* Unwilling to be randomized
* Unwilling to continuously wear and regularly sync/charge the Fitbit device during the study period.
* Unable to read and speak in English
* Unwilling to provide written informed consent to participate
* Cognitive impairment (score <21 on the TICS-M) prior to baseline assessment
* History of stroke, transient ischemic attack, other neurological disorders, or brain surgery involving tissue removal

Min Age: 21 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2021-01-15 (Actual); Primary Completion 2022-07-07 (Actual); Study Completion 2022-07-07 (Actual)

PRIMARY OUTCOMES:
intervention attendance | 1 month post-chemotherapy
  completion of telecoaching sessions
Participant satisfaction: survey | 1 month post-chemotherapy
  usability survey
recruitment yield | Baseline
  number of women who enroll compared to the number of contacts of eligible women required to obtain target sample size
retention | 1 month post-chemotherapy
  proportion of participants providing post-intervention data
acceptability of intervention: in-depth interview | 1 month post-chemotherapy
  in-depth interview to gather participant perceptions on the acceptability and usefulness of the mobile app features

SECONDARY OUTCOMES:
Change in Stroop task performance | Baseline, 1 month post-chemotherapy
  Interference score on Stroop task
Change in Task-Switch task performance | Baseline, 1 month post-chemotherapy
  Reaction time on Task-Switch
Change in Trails task performance | Baseline, 1 month post-chemotherapy
  Completion time of Trails
Change in N-Back task performance | Baseline, 1 month post-chemotherapy
  Correct responses on N-back
Change in Spatial Working Memory task performance | Baseline, 1 month post-chemotherapy
  Correct responses on Spatial Working Memory task
Change in Auditory Verbal Learning Task (AVLT) performance | Baseline, 1 month post-chemotherapy
  Total numbered recalled on AVLT
Change in objective physical activity behavior | Baseline, 1 month post-chemotherapy
  Objective activity behavior (average minutes of physical activity per day) will be measured using actigraphy.

OTHER OUTCOMES:
Change in cancer-related Fatigue | Baseline, 1 month post-chemotherapy
  The Functional Assessment in Chronic Illness Therapy (FACIT) - Fatigue Scale will be used to measure cancer-related fatigue. Scores range from 0-52, with higher scores indicating less cancer-related fatigue.
Momentary symptoms | 14 days 4 times per day at each of the following time points: baseline, mid-intervention (2-3 months from baseline), 1 month post-chemotherapy
  A brief ecological momentary assessment prompted to participants' smartphones will be used to measure momentary symptoms, including anxiety, stress, fatigue, focus, pain, and nausea.

CONTACTS AND LOCATIONS:
Overall Officials: Laura D Bilek, PT, PhD, Principal Investigator — University of Nebraska
Locations (1):
- University of Nebraska Medical Center, Omaha, Nebraska, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data will be available to other researchers upon request and approval by the PI.
Supporting Information: Study Protocol, CSR
Time Frame: After primary manuscripts have been published.
Access Criteria: To be determined upon research request.

DOCUMENTS (1):
  • Informed Consent Form (2021-10-07): https://cdn.clinicaltrials.gov/large-docs/87/NCT04562987/ICF_000.pdf